CLINICAL TRIAL: NCT07160023
Title: Local Registry of Primary Cutaneous T-cell Lymphomas
Acronym: CuTLy
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Valeria Brazzelli, Principal Investtigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: CuTLy
Record Dates: First submitted 2025-02-17; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-02

CONDITIONS: Primary Cutaneous T-cell Lymphomas NCT Number

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with primary cutaneous T-cell lymphoma: Patients with primary cutaneous T-cell lymphoma attending the Dermatology Unit Outpatient Clinics

SUMMARY:
This registry aims to collect retrospective and prospective data on patients with primary cutaneous T-cell lymphoma who are treated at the Dermatology Clinic of the IRCCS Policlinico San Matteo Foundation.

ELIGIBILITY:
Inclusion criteria:

* primary cutaneous T-cell lymphoma attending the outpatient clinics of the Dermatology Unit in Pavia

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with primary cutaneous T-cell lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2033-10-12 (Estimated); Study Completion 2033-10-12 (Estimated)

PRIMARY OUTCOMES:
prevalence of cutaneous T-cell lymphoma (CTCL) variants | October 2033
  The prevalence and the exact binomial 95% CI will be presented.

SECONDARY OUTCOMES:
survival among the various subtypes of CTCL | October 2033
  To compare survival among the various subtypes of CTCL, the survival rate will be reported as deaths per 100 person-years; the start date of follow-up will be the diagnosis of the disease. The groups will be compared using the log-rank test and survival will be described using Kaplan-Meier curves.
Association between clinical, histopathological and immunophenotypic characteristics of patients with cutaneous T-cell lymphoma and overall survival | October 2033
  A Cox model will be used to derive the hazard ratio (HR) and relative 95% CI. Harrell's c statistic will be calculated for the model's ability to discriminate. Estimates will be adjusted as far as possible for potential confounding factors.
dermatoscopic features of cutaneous T-cell lymphomas | October 2033
  Descriptive statistics will be calculated for each type of cutaneous lymphoma.

CONTACTS AND LOCATIONS:
Locations (1):
- SC Dermatologia, Fondazione IRCCS Policlinico San Matteo, Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No